CLINICAL TRIAL: NCT03359668
Title: CT Detection of Metastatic Lymphadenopathy in Papillary Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11-0192-C
Record Dates: First submitted 2017-11-16; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Intervention Model Description: Each patient had CT imaging with and without IV contrast
Who Masked: Investigator
Masking Description: The investigator will read the randomized non-contrast CTs separately from the contrast-enhanced CTs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-contrast-enhanced CT (Experimental): Comparison of non-contrast CT to the standard-of-care contrast-enhanced CT of the head and neck in detection of suspicious lymph nodes
  Interventions: Diagnostic Test: Use of IV contrast during head and neck CT
- Contrast-enhanced CT (Active Comparator): Comparison of non-contrast CT to the standard-of-care contrast-enhanced CT of the head and neck in detection of suspicious lymph nodes
  Interventions: Diagnostic Test: Use of IV contrast during head and neck CT

INTERVENTIONS:
Diagnostic Test: Use of IV contrast during head and neck CT — Use of IV contrast during head and neck CT
  Other Names: Non-contrast-enhanced CT of the head and neck

SUMMARY:
Localized thyroid cancer is potentially curable. Before thyroid surgery, an ultrasound test is done to see if cancer has spread to the lymph nodes in the neck. Excellent for evaluation of the thyroid gland, this test has limitations in evaluating larger anatomic areas, like all groups of lymph nodes in the neck. It has a limited area of coverage making it difficult to define an area of interest, depends on the skill level of the person performing it, and is difficult to exactly reproduce on follow-up. For these reasons, CT is often performed in these patients but without intravenous (IV) contrast since iodine-based contrast agents may saturate the thyroid, limiting the usefulness of other iodine-based diagnostic and treatment options. However, contrast-CT can give more detailed information about tumor spread including spread to lymph nodes. We aim to determine if use of IV contrast agent during CT leads to earlier and more accurate detection of lymph node disease from thyroid cancer.

DETAILED DESCRIPTION:
Papillary thyroid cancer represents 75% of all epithelial thyroid malignancies. Imaging not only delineates the primary tumour within the thyroid gland, but also helps assess lymph nodal metastatic disease helping guide the extent of surgical neck dissection. Ultrasonography (US) is the current imaging standard (American Thyroid Association guidelines). However, US is limited by operator skills and lacks specific anatomic references essential to plan surgery. CT is performed to address these issues, often without intravenous (IV) contrast for fear of saturating thyroid tissue with iodine present in it, thus rendering iodine-labeled nuclear testing/treatment ineffective for a finite period of time. But post-contrast nodal enhancement is a predominant morphologic feature of suspicious lymphadenopathy in papillary thyroid cancer, and contrast-CT can facilitate an earlier detection. Iodine-saturation is not a concern in these patients as its concentration will normalize during recovery.

In pre-surgical thyroidectomy patients with proven papillary thyroid cancer, the use of intravenous (IV) CT contrast improves the reliability and accuracy of suspicious head and neck lymph node detection, in comparison to CT without IV contrast.

This study will help define the accuracy and reliability of intravenous (IV) contrast use in the detection of metastatic neck lymph nodes from papillary thyroid cancer. Improved detection of suspicious metastatic lymphadenopathy in papillary thyroid cancer will directly impact the patient's management since the surgical plan will be based upon the detection of these suspicious lymph nodes. CT imaging provides an anatomically relevant approach to surgery and is consistently reproducible, thus providing direct benefits to the pre-surgical assessment. Ultimately, this will result in decreased nodal recurrences within the neck.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative thyroidectomy patients with pathology-proven papillary thyroid cancer (PTC) needing lymph node staging for potential neck dissection.

Exclusion Criteria:

* Patients with history of prior surgery within the head and neck.
* Patients with history of prior radiation to the head and neck.
* Patients with history of lymphoma, leukemia, or other lymphoproliferative disorders affecting the head and neck.
* Pregnant/breast feeding patients (by question).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Increased detection of suspicious lymph nodes in PTC with IV-contrast enhanced CT | up to 7 years

IPD SHARING:
Plan to Share IPD: No